CLINICAL TRIAL: NCT05383716
Title: A Prospective, Single-arm PhaseⅡTrial of Neoadjuvant/Adjuvant Pembrolizumab Plus Platinum-doublet Chemotherapy (Chemo) in IIa-IIIb NSCLC
Brief Title: Neoadjuvant/Adjuvant Pembrolizumab Plus Chemotherapy
Acronym: NeoP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wang mengzhao, Prof., Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-2847
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Non Small Cell Lung Cancer; Neoadjuvant Therapy; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemotherapy plus pembrolizumab (Experimental): Two to four cycles of neoadjuvant chemotherapy in combination with pembrolizumab will be administered before surgery, followed by another one to two cycles of chemotherapy plus pembrolizumab after surgery (4 cycles neoadjuvant/adjuvant chemotherapy in total ) then use pembrolizumab monotherapy for up to 1 year
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Two to four cycles of neoadjuvant chemotherapy in combination with pembrolizumab will be administered before surgery, followed by another one to two cycles of chemotherapy plus pembrolizumab after surgery (4 cycles neoadjuvant/adjuvant chemotherapy in total ) then use pembrolizumab monotherapy for up to 1 year.
  Other Names: Keytruda

SUMMARY:
A phase II, single-arm, open-label study evaluating feasibility, safety and efficacy of combined chemotherapy and pembrolizumab as neoadjuvant/adjuvant therapy in stage IIa-IIIB NSCLC adult patients followed by adjuvant PD-(L)1 inhibitor treatment for up to 1 year

DETAILED DESCRIPTION:
Two to four cycles of neoadjuvant chemotherapy in combination with pembrolizumab will be administered before surgery, followed by another one to two cycles of chemotherapy plus pembrolizumab after surgery (4 cycles neoadjuvant/adjuvant chemotherapy in total ) then use pembrolizumab monotherapy for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Primary non-small cell lung cancer (NSCLC) confirmed by cytology or histology
2. Stage IIa to selected IIIb ( t1-4, n0-2 ) NSCLC according to the TNM stage (8th Edition) of IASLC, which is considered to be resectable;
3. At least one evaluable focus judged according to RECIST 1.1 standard (on spiral CT, the longest diameter of tumor should be at least 10 mm, the shortest diameter of metastasis lymphnode should be at least 20 mm)
4. ECOG PS 0 or 1
5. Adequate tumor samples available for gene detection (EGFR/ALK /ros1) with non-squamous and specimens for PD-L1 immunohistochemistry (IHC) in all the subjects.
6. Male or female, ≥ 18 years old
7. Adequate blood function: absolute neutrophil count (ANC) ≥ 2 × 109 / L, platelet count ≥ 100 × 109 / L and hemoglobin 110 ≥ 9 g / dl
8. Adequate liver function: total bilirubin ≤ upper limit of normal value (ULN); AST and alt ≤ upper limit of normal value (ULN); alkaline phosphatase ≤ upper limit of normal value (ULN)
9. Adequate renal function: serum creatinine ≤ upper limit of normal value (ULN) or calculated creatinine clearance ≥ 60ml / min
10. No history of using anti-tumor drug treatment before
11. For patients who have had previous surgery, it is required that more than 4 weeks have passed since the start of study treatment, and the patients have recovered
12. Sign the informed consent form (the informed consent form needs to be approved by the independent ethics committee, and the informed consent of the patient should be obtained before starting any substantive trial procedure)

Exclusion Criteria:

1. Carrying activating mutations in the TK domain of EGFR or any variety of alterations in the ALK gene or other known targetable driver mutations.
2. Active, known or suspected autoimmune disease.
3. Other active malignancy in the last 5 years (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast).
4. Prior treatment with anti-PD-1, anti-CTLA-4 (cytotoxic T lymphocyte-associated antigen (CTLA-4), or anti-PD-L1 therapeutic antibody or pathway-targeting agents
5. History of allergy to study drug components excipients
6. Having any uncontrolled systemic diseases, including active infection, uncontrolled hypertension, diabetes, unstable angina, congestive heart failure, acte myocardial infarction (within 3 months before treatment), serious arrhythmia requiring drug treatment, liver, kidney and metabolic diseases
7. Women in pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
MPR(major pathologic response) | Up to 8weeks
  more than 90 percent decrease in viable tumor

SECONDARY OUTCOMES:
Complete pathological (CPR) response rate | 8 weeks
  The investigator assessed CPR rate was defined as the percentage of subjects who achieved complete pathological remission (no residual tumor in lung and lymph nodes)
EFS (event free survival) | 8 weeks
  the time length from randomization (mainly from the receipt of pathology and genetic diagnosis reports)to any of the following events: disease progression, disease recurrence or death from any cause. Disease progression or relapse will be assessed according to RECIST 1.1
OS (overall survival) | 8 weeks
  the time length from randomization (mainly from the receipt of pathology and genetic diagnosis reports)to death from any cause.
Incidence of adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 8 weeks
  Evaluate adverse events of any cause, treatment-related adverse events, immune-mediated adverse events according to NCI-CTCAE V5.0
Evaluate tissue biomarkers | 8 weeks
  The goals for these analyses are for hypothesis generating. The results will need to be confirmed by future studies.
  Used for hypothesis generating. Transcriptome analysis identity markers with efficacy and/or toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, MD., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The result of the study and all the supporting informations will be shared in the form of publishing article.